CLINICAL TRIAL: NCT05997875
Title: Transforming Hemodialysis-Related Vascular Access Education (THRiVE)
Brief Title: Transforming Hemodialysis-Related Vascular Access Education
Acronym: THRiVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Laura Dember, MD, Professor of Medicine and Epidemiology, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 853978
Record Dates: First submitted 2023-07-19; First posted 2023-08-18 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Disease; Hemodialysis Vascular Access
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Education (Experimental)
  Interventions: Behavioral: Educational Materials; Behavioral: Usual Care; Other: Patient Lists for Clinicians: System-Level Intervention
- Education-Plus (Experimental)
  Interventions: Behavioral: Educational Materials; Behavioral: Motivational Interviewing; Behavioral: Usual Care; Other: Patient Lists for Clinicians: System-Level Intervention
- Usual Care (Other)
  Interventions: Behavioral: Usual Care; Other: Patient Lists for Clinicians: System-Level Intervention

INTERVENTIONS:
Behavioral: Educational Materials — Participants are provided with the "Getting Ready: Your Vascular Access Journey" video and brochure about hemodialysis vascular access. The video is available for viewing via smartphone or computer. Both the brochure and video were created with input from patients with chronic kidney disease.
  Arms: Education; Education-Plus
Behavioral: Motivational Interviewing — Participants receive coaching with telehealth-based motivational interviewing designed to prepare participants to move forward with vascular access creation. Motivational interviewing will consist of a minimum of 3 and maximum of 8 telehealth sessions with a coach. The coach will use patient-centered communication skills to work though the stages of pre-contemplative, contemplative, preparation, action, and maintenance of an arteriovenous vascular access.
  Arms: Education-Plus
Behavioral: Usual Care — Participants receive the non-standardized vascular access counseling and referral to the chronic kidney disease education class that comprises the standard care provided by their nephrology clinic.
Other: Patient Lists for Clinicians: System-Level Intervention — Nephrologists and clinic staff receive monthly, provider-specific, lists of patients potentially appropriate for AV access planning based on eGFR thresholds and kidney failure risk. These criteria identify patients at risk for progression to dialysis and are congruent with evidence-based guidelines for optimal timing of AV access evaluation referral.

SUMMARY:
The focus of this study is on vascular access for hemodialysis. This is a randomized clinical trial testing 3 educational approaches to help patients with advanced chronic kidney disease prepare for placement of hemodialysis vascular access. Study participants will each be assigned to one of the 3 approaches: 1) "Education", in which participants will be given a video and brochure that provide information about the types of vascular access and what can be expected before and after the vascular access is placed, 2) "Education-Plus", in which participants will be given the video and brochure and will also have sessions by telehealth with a motivational interviewing coach to provide additional support around vascular access placement, and 3) "Usual Care", in which participants will have the usual education provided by their kidney doctor and clinic staff just as if they were not in the study. Participants in all 3 groups will be asked to complete questionnaires by telephone and may be invited to be interviewed about their experience with the study intervention at the end of the study. Study participation will last for about 12 months, with most of the study activities taking place during the first 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Nephrology visit for chronic kidney disease during the last 18 months
3. Most recent eGFR less than or equal to 20 ml/min/1.73 m2 or 2-year Kidney Failure Risk Equation score greater than 40%
4. Documentation in the medical record or confirmation from the treating nephrologist of a patient-nephrologist discussion about hemodialysis

Exclusion Criteria:

1. Planning for peritoneal dialysis, preemptive transplant, or conservative management of kidney failure
2. Previous placement of an AV access
3. Prior appointment with surgeon for AV access evaluation or creation
4. Cognitive dysfunction or severe visual impairment that prevents use of the education materials
5. Does not speak either English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Surgery for Creation of Hemodialysis Arteriovenous Access (Effectiveness outcome) | Within 12 months after randomization or before hemodialysis initiation, whichever comes first
  The proportion of participants who have arteriovenous access creation surgery.

SECONDARY OUTCOMES:
Scheduled Appointment with Surgeon for Vascular Access Evaluation (Effectiveness outcome) | Within 12 months after randomization or before hemodialysis initiation, whichever comes first
  The proportion of participants with a scheduled appointment with a surgeon for evaluation for vascular access creation.
Completed Appointment with Surgeon for Vascular Access Evaluation (Effectiveness outcome) | Within 12 months after randomization or before hemodialysis initiation, whichever comes first
  The proportion of participants with a completed appointment with a surgeon for evaluation for vascular access creation.
Imaging for Planning Arteriovenous Vascular Access Creation (Effectiveness outcome) | Within 12 months after randomization or before hemodialysis initiation, whichever comes first
  The proportion of participants with completed vascular imaging via ultrasound or angiography for planning arteriovenous vascular access creation surgery.
Usable Arteriovenous Vascular Access (Effectiveness outcome) | Up to 4 years after randomization (full duration of the trial)
  For participants who start hemodialysis, the proportion with a usable arteriovenous access at dialysis initiation.
Vascular Access Knowledge (Effectiveness outcome) | 12 weeks after randomization
  The change from baseline in vascular access knowledge as measured by the Patient Perceived Vascular Access Knowledge scale. The total score ranges from 0 to 10, with higher scores indicating a higher level of vascular access knowledge.
Decision Self-Efficacy (Effectiveness outcome) | 12 weeks after randomization
  The change from baseline in decision self-efficacy as measured by the Decision Self-Efficacy Scale. The total score ranges from 0 to 11, with higher scores indicating a higher level of self-efficacy when making decisions about hemodialysis vascular access.
Preparedness for Decision-Making (Effectiveness outcome) | 12 weeks after randomization
  A participant's level of preparedness for decision-making as measured by the Preparation for Decision-Making Scale. The total score ranges from 0-100, with higher scores indicating a higher perceived level of preparation for decision-making.
Characteristics of Eligible Patients - quantitative reach assessment (Implementation outcome) | Pre-Enrollment
  An assessment of the demographic and socioeconomic characteristics of patients who are eligible for the trial.
Characteristics of Enrolled Participants - quantitative reach assessment (Implementation outcome) | Baseline
  An assessment of the demographic and socioeconomic characteristics of patients who enroll in the trial.
Characteristics of Participants who Complete the Trial - quantitative reach assessment (Implementation outcome) | 12 months
  An assessment of the demographic and socioeconomic characteristics of participants who complete the trial.
Characteristics of Participants who Withdraw from the Trial - quantitative reach assessment (Implementation outcome) | From eligibility until 12 months
  An assessment of the demographic and socioeconomic characteristics of participants who withdraw from the trial.
Declined Enrollment - quantitative reach assessment (Implementation outcome) | Pre-enrollment
  The reasons for declining enrollment as documented in screening logs and provided in aggregate for an enrolling center.
Reasons for Participation - qualitative reach assessment (Implementation outcome) | 12-16 weeks after randomization
  The reasons for participation and non-participation as identified through qualitative interviews
Reasons Nephrologists Opt-Out on Behalf of Patients - qualitative reach assessment (Implementation outcome) | Up to 4 years after trial initiation (full duration of the trial)
  The reasons that nephrologists opt out of having an eligible patient approached by the research team for possible enrollment as identified through qualitative interviews.
Acceptability Intervention Measure - quantitative acceptability assessment (Implementation outcome) | 12 -16 weeks after randomization
  The acceptability of the intervention as measured by the Acceptability of Intervention Measure (AIM). The total score ranges from 1-5, with higher scores indicating a higher level of acceptability of the intervention.
Acceptability of Intervention Content, Delivery, and Accessibility - qualitative acceptability assessment (Implementation outcome) | 12 to 16 weeks after randomization
  The acceptability of the content, delivery, and accessibility of educational materials and motivational interviewing coaching as identified through qualitative interviews.
Chronic Kidney Disease Class Attendance - quantitative fidelity assessment (Implementation outcome) | Within 12 months
  The proportion of participants who attend a Chronic Kidney Disease education class provided by their nephrology clinic
Receipt of Educational Materials - quantitative fidelity assessment (Implementation outcome) | Within 12 weeks after randomization
  The proportion of participants with confirmed receipt of the "Getting Ready" brochure (only be assessed for the Education and Education-Plus groups)
Viewing of Video - quantitative fidelity assessment (Implementation outcome) | Within 12 weeks after randomization
  The proportion of participants with confirmed viewing of the "Getting Ready" video, which will only be assessed for the Education and Education-Plus groups.
Completed Motivational Interviewing Sessions - quantitative fidelity assessment (Implementation outcome) | Within 12 months after randomization
  The proportion of participants who completed the scheduled motivational interviewing sessions (only be assessed for the Education-Plus group)
Brochure Delivery Mode - quantitative barriers/facilitators assessment (Implementation outcome) | Within 12 weeks after randomization
  The selected mode for delivery of the "Getting Ready" brochure by center, clinic, and participant sociodemographic characteristics.
Video Delivery Mode - quantitative barriers/facilitators assessment (Implementation outcome) | Within 12 weeks after randomization
  The selected mode for viewing of the "Getting Ready" video by center, clinic, and participant sociodemographic characteristics.
Participant Contact Attempts for Motivational Interviewing - quantitative barriers/facilitators assessment (Implementation outcome) | 12 month period after randomization
  The number and type (email, phone, text messaging) of attempted and confirmed participant contacts by the motivational interviewing coach.
Missed Motivational Interviewing Sessions - quantitative barriers/facilitators assessment (Implementation outcome) | 12 month period after randomization
  The number of missed motivational interviewing sessions.
System-Level Barriers to Arteriovenous Access Creation From Clinical Staff Perspective - qualitative implementation/barriers assessment (Implementation outcome) | Up to 4 years after trial initiation (full duration of the trial)
  System-level barriers to arteriovenous vascular access creation and relevant system contextual factors as identified through qualitative interviews.
System-Level Barriers to Arteriovenous Access Creation From Participant Perspective - qualitative implementation/barriers assessment (Implementation outcome) | Within 12 months
  System-level barriers to arteriovenous vascular access creation and relevant system contextual factors as identified through qualitative interviews.

OTHER OUTCOMES:
Creation of Arteriovenous Vascular Access Without Subsequent Need for Hemodialysis | Up to 4 years after randomization (full duration of the trial)
  The creation of an arteriovenous vascular access without a subsequent need for hemodialysis is a potential unintended consequence of interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Laura M. Dember, MD, Principal Investigator — University of Pennsylvania; Jennifer E. Flythe, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill; Deidra Crews, MD, ScM, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania